CLINICAL TRIAL: NCT06984302
Title: HYPOTENSION PREDICTION INDEX FOR HEMODYNAMIC OPTIMIZATION IN MAJOR VASCULAR SURGERY
Brief Title: A PREDICTIVE ALGORITHM IN AORTIC SURGERY
Acronym: HYVAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7458
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proactive group (Experimental): in this group patients will be managed by a predictive hemodynamic algorithm
  Interventions: Other: proactive therapy
- control group (No Intervention): drugs and fluids will be given based on mean arterial pressure and stroke volume variation respectively

INTERVENTIONS:
Other: proactive therapy — drugs and fluids will be given based on the hypotension prediction index
  Arms: proactive group

SUMMARY:
We will enroll patients scheduled for abdominal aortic aneurysm repair and divide in two groups; in the control group the hemodynamic optimization will be made based on standard cardiovascular parameters showed in the Hemosphere platform. In the interventional group the hemodynamic optimization will be made based on the hypotension prediction index.

ELIGIBILITY:
Inclusion Criteria:

* planned aortic surgery acceptance of written informed consent

Exclusion Criteria:

* body mass index > 35 kg/m2
* atrial fibrillation
* urgent surgery
* end-stage renal disease
* pregnancy
* refusal of the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
time weighted average of mean arterial presure under 65 mmHg | at the end of surgery
  we will assess the magnitude of intraoperative arterial hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy